CLINICAL TRIAL: NCT04762329
Title: Manage My Pain at Chronic Pain Clinics in Urban, Community, and Rural Hospitals
Brief Title: Manage My Pain at Chronic Pain Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Centres of Excellence (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-6201
Record Dates: First submitted 2020-10-26; First posted 2021-02-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Pain; Psychology; Patient Oriented Research; Quality of Life; Digital Health; Chronic Pain; Pain App; Virtual Care; mHealth; Pain Management; Chronic Disease Management; Remote Monitoring
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia | interventions — Matrix Metalloproteinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group using Manage My Pain (MMP) digital application for pain data (Experimental): Participants completed pain related questionnaires on the following pain related outcomes - anxiety, depression, catastrophizing, disability, patient impression of change, and daily opioid consumption at baseline on initial visit and as a part of the first follow-up clinical visits, on the Manage My Pain (MMP) digital application
  Interventions: Other: Manage My Pain (MMP) digital pain app group
- Patient group using paper format for pain data (No Intervention): Participants completed pain related questionnaires on the following pain related outcomes - anxiety, depression, catastrophizing, disability, patient impression of change, and daily opioid consumption at baseline on initial visit and as a part of the first follow-up clinical visits on paper format or phone interviews.

INTERVENTIONS:
Other: Manage My Pain (MMP) digital pain app group — To evaluate the extent of patient engagement with the Manage My Pain (MMP) digital application when used in a clinical setting
  Arms: Patient group using Manage My Pain (MMP) digital application for pain data

SUMMARY:
The overall objective of this Early Adoption project is to gather evidence for how Managing My Pain Program (MMP), a novel digital pain management application can enable better care at home for chronic pain sufferers in the province of Ontario, Canada across 4 sites in urban, community, and rural settings

DETAILED DESCRIPTION:
Chronic pain imposes a large burden on individuals and society. A patient-centric digital chronic pain management application, Managing My Pain Program (MMP) that incorporates validated questionnaires can be used to enhance communication between providers and patients and promote self-management to evaluate the extent of patient engagement with the app when used in clinical settings.

The main objectives for this project is to evaluate the engagement in patients using MMP, and to assess improvements in clinical outcomes directly relevant for pain management, as measured by clinically-validated tools.

ELIGIBILITY:
Inclusion Criteria:

* New patients with chronic pain conditions referred to participating sites with pain programs to adopt the MMP tool into clinical practice.

Exclusion Criteria:

* Patients declining to consent for the study
* Patients withdrawing from the study at a later time after consenting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Evaluating engagement based on adoption and retention rates | 24 months
  Evaluating the number of patients who elected to use the Manage My Pain (MMP) application, and determining how long they used the app in the short-term (4.5 months) and long-term (4.5-7 months) follow-ups

SECONDARY OUTCOMES:
Change in depression as measured by the Patient Health Questionnaire 9-item (PHQ-9) | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum score of 0, maximum score of 27. The higher the score, the higher the severity of depression.
Change in anxiety as measured by the General Anxiety Disorder 7-item Questionnaire (GAD-7) | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum score of 0, maximum score of 21. The higher the score, the higher the severity of anxiety.
Change in pain disability as measured by the Pain Disability Index (PDI) | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum score of 0, maximum score of 70. The higher the score, the higher the severity of pain disability.
Change in pain catastrophizing and measured by the Pain Catastrophizing Scale (PCS) | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum score of 0, maximum score of 52. The higher the score, the higher the severity of pain catastrophizing.
Change in opioid consumption as measured by Oral Morphine Equivalents (OME) | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum amount of 0, no maximum amount. The higher the amount the more opioid they are taking
Change in patient satisfaction as measured by the Patient Global Impression of Change (PGIC) scale | Short-term (4.5 months) and long-term (4.5-7 months)
  Minimum score of 1, maximum score of 7. The higher the score, the higher the level of patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD was collected during the study to share

REFERENCES:
- [Background] Portelli P, Eldred C. A quality review of smartphone applications for the management of pain. Br J Pain. 2016 Aug;10(3):135-40. doi: 10.1177/2049463716638700. Epub 2016 Apr 19. PMID 27583140
- [Background] Alexander JC, Joshi GP. Smartphone applications for chronic pain management: a critical appraisal. J Pain Res. 2016 Sep 26;9:731-734. doi: 10.2147/JPR.S119966. eCollection 2016. No abstract available. PMID 27713649
- [Background] Salazar A, de Sola H, Failde I, Moral-Munoz JA. Measuring the Quality of Mobile Apps for the Management of Pain: Systematic Search and Evaluation Using the Mobile App Rating Scale. JMIR Mhealth Uhealth. 2018 Oct 25;6(10):e10718. doi: 10.2196/10718. PMID 30361196
- [Derived] Bhatia A, Kara J, Janmohamed T, Prabhu A, Lebovic G, Katz J, Clarke H. User Engagement and Clinical Impact of the Manage My Pain App in Patients With Chronic Pain: A Real-World, Multi-site Trial. JMIR Mhealth Uhealth. 2021 Mar 4;9(3):e26528. doi: 10.2196/26528. PMID 33661130